CLINICAL TRIAL: NCT07094516
Title: A Randomized, Placebo-controlled, Parallel Group, 72-week Study to Evaluate the Efficacy and Safety of VHB937 in Participants With Early Alzheimer's Disease Followed by an Extension
Brief Title: A Clinical Trial to Learn About the Effects of VHB937 in People With Early Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVHB937A12201
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; AD; Dementia; Monoclonal Antibody
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Double-blind, Randomized
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded placebo for infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VHB937 Low Dose (Experimental): I.V. infusions
  Interventions: Biological: VHB937
- VHB937 High Dose (Experimental): I.V. infusions
  Interventions: Biological: VHB937
- Placebo (Placebo Comparator): I.V. infusions
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VHB937 — VHB937 solution for infusion
  Arms: VHB937 Low Dose
Biological: VHB937 — VHB937 solution for infusion
  Arms: VHB937 High Dose
Other: Placebo — Solution for infusion
  Arms: Placebo

SUMMARY:
This is a multicentre, randomized, double-blind, placebo-controlled, parallel group Phase II study to evaluate the efficacy and safety of VHB937 in participants with early AD followed by an Extension. The double-blind part is 72 weeks long, followed by an extension.

DETAILED DESCRIPTION:
The purpose of this study is to find out whether treatment with VHB937 is safe and beneficial in people with early Alzheimer's disease. The study will evaluate the safety of VHB937, as well as its effects on memory and other thinking abilities, on daily activities, and on changes in the brain. The study will also observe and measure how VHB937 is processed by the body and how the body responds to it.

ELIGIBILITY:
Key Inclusion Criteria

* Male or female participants 50 to 85 years of age
* Diagnosis of Mild Cognitive Impairment (MCI) due to AD or mild AD
* Clinical Dementia Rating (CDR) Global score of 0.5 or 1.0
* Confirmation of AD based on cerebral spinal fluid (CSF) biomarkers or amyloid PET imaging
* Reliable study partner who can accompany the participant at study visits
* If on symptomatic AD treatment (AChEIs/memantine), on a stable dose prior to starting study treatment

Key Exclusion Criteria

* Dementia due to a condition other than AD, including but not limited to, frontal temporal dementia, Parkinson's disease, dementia with Lewy bodies, Huntington disease, vascular dementia.
* History or current diagnosis of cardiac conditions or ECG abnormalities indicating significant risk of safety for participants in the study
* Transient ischemic attacks (TIA) or stroke occurring within 12 months
* Clinical evidence of liver or renal disease/injury
* Current major depressive episode that is not adequately controlled, history of schizophrenia, other chronic psychosis
* Significant neurological disease other than dementia (e.g. serious brain infection, traumatic brain injury, multiple concussions, epilepsy or recurrent seizures
* Presence of suicidal ideation within 6 months or suicidal behavior within 2 years before Screening
* Presence of cancer, HIV, Hep B, Hep C, uncontrolled thyroid disease, uncontrolled diabetes
* Taking any prohibited medications

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2028-09-14 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Clinical Dementia Rating scale - Sum of Boxes (CDR-SB) | Baseline and Week 72
  The CDR is a measure of cognition and function, widely used in clinical research in AD. The scale assesses six domains: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. Based on in-depth semi-structured interview, each domain is assigned a score, which is summed to obtain the Sum of Boxes (SB) score, ranging from 0 to 18 with higher scores indicating worse condition

SECONDARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From First treatment to end of study (up to 63 months approximately)
  Incidence and severity of AEs and SAEs by treatment group, including Safety findings, Laboratory tests, Vital signs and, ECG findings qualifying and reported as AEs.
Change from Baseline in Clinical Dementia Rating scale - Sum of Boxes (CDR-SB) | Baseline over time until Week 72
  The CDR is a measure of cognition and function, widely used in clinical research in AD. The scale assesses six domains: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care.
Change from Baseline in Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog14) | Baseline over time until Week 72
  The ADAS-Cog is is a 14-item clinical assessment tool to measure cognition. The ADAS-Cog14 score ranges between 0 and 90, with higher scores indicating worse cognitive performance
Change from Baseline in instrumental activities of daily living (iADL) on the Alzheimers Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) scale | Baseline over time until Week 72
  The ADCS-ADL is a 23-item study partner scale designed to assess the ability of patients with AD to carry out basic activities of daily living (bADLs) and instrumental activities of daily living (iADLs). For each item, the study partner is asked whether the participant attempted the activity in the 4 preceding weeks. Where 'yes' is the answer, the study partner is asked to rate the patient's level of performance according to a set of descriptors tailored to that activity. Scores on iADL sub-scale range between 0 and 59, with lower scores reflecting greater disease severity
Pharmacokinetic parameters of VHB937 in serum - Cmax | Baseline over time until Week 72
  Cmax - The maximum concentration of VHB937 in serum
Pharmacokinetic parameters of VHB937 in serum - Tmax | Baseline over time until Week 72
  Tmax - The time to reach the maximum concentration of VHB937 in serum
Pharmacokinetic parameters of VHB937 in serum - Ctrough | Baseline over time until Week 72
  Ctrough - Minimum observed concentration of VHB937 in CSF
VHB937 immunogenicity in serum | Baseline over time until Week 72
  Determination of anti-VHB937 antibodies in serum at selected timepoints

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Jem Research Institute, Atlantis, Florida
  - Visionary Investigators Network, Aventura, Florida
  - K2 Medical Research LLC, Maitland, Florida
  - Charter Research The Villages, The Villages, Florida
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Abington Neurological Associates Ltd, Willow Grove, Pennsylvania
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.